CLINICAL TRIAL: NCT06787326
Title: Effect of the BioFire FilmArray (BCID2) for the Rapid Detection of Bloodstream Infection in Haematologic Patients With Febrile Neutropenia (ONFIRE Study): Study Protocol of a Prospective, Multicentre Observational Study
Brief Title: Effect of the BioFire FilmArray (BCID2) for the Rapid Detection of Bloodstream Infection in Haematologic Patients With Febrile Neutropenia
Acronym: ONFIRE
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Carlota Gudiol, Professor, MD, PhD, Hospital Universitari de Bellvitge
Other Study IDs: ICPS029/22; PI21/01280 (Other Grant/Funding Number: Instituto de Salud Carlos III)
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Haematological Malignancy; Febrile Neutropenia; Blood Stream Infection
Keywords: Blood Stream Infection; Bacteraemia; Febrile Neutropenia; BioFire FilmArray (BCID2); Haematologic Malignancy; Neutropenic Cancer Patients
MeSH Terms: conditions — Hematologic Neoplasms; Febrile Neutropenia; Toxemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to assess if the molecular diagnostic tool BioFire FilmArray BCID2 is more useful for the microbiological diagnosis of bloodstream infections in hematological patients with febrile neutropenia, compared to the conventional microbiologic studies.

The study compares the sensibility and specificity of these two techniques.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients hospitalised for the treatment of haematological malignancy or undergoing an autologous or allogeneic hematopoietic stem cell transplant or receiving CAR-T cell therapy
* Patients presenting with febrile neutropenia (defined as axillary temperature ≥ 38.0°C and <500 neutrophils/mm3 or <1000 with an expected rapid decrease in 24-48 hours),
* Patient to whom blood cultures are ordered as standard care for the microbiological diagnosis of the febrile neutropenia episode.

Exclusion Criteria:

* Axillary temperature <37.5ºC.
* High clinical suspicion of a non-infectious cause of fever at the moment when blood cultures are drawn (high suspicion of drug related fever, infusion reaction).
* Previously enrolled patients in whom the time between inclusion and the current episode is less than four weeks.
* Patients with febrile neutropenia in whom no blood cultures are drawn.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult patients (age ≥18 years) hospitalised for the treatment of leukaemia, lymphoproliferative syndrome, myelodysplastic syndrome, multiple myeloma, medullary aplasia, or patients undergoing an autologous or allogeneic hematopoietic stem cell transplant or receiving CAR-T cell therapy, who develop febrile neutropenia (defined as axillary temperature ≥ 38.0°C and <500 neutrophils/mm3 or <1000 with an expected rapid decrease in 24-48 hours), and who have diagnostic blood cultures ordered as standard care for the microbiological diagnosis of the febrile neutropenia episode.
Sampling Method: Probability Sample
Enrollment: 228 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of BioFire FilmArray BCID2 panel compared to conventional blood cultures. | 14 days
  For the analysis of the primary endpoint:
  * The sensitivity (proportion of positive results) of the BioFire FilmArray BCID2 panel will be compared with the sensitivity of the companion blood cultures. The results of the BioFire FilmArray samples that meet the definitions of "Proven bloodstream infection", "Probable bloodstream infection" and "Possible bloodstream infection" will be considered as positive results. The results will be assessed at Day 14 from the sample collection. The positive predictive value of both techniques will be calculated and compared.
  * The specificity (proportion of negative results) of the FilmArray BCID2 panel will be compared with the specificity of the companion blood cultures. The results will be assessed at Day 14 from the sample collection. The negative predictive value of both techniques will be calculated and compared.

SECONDARY OUTCOMES:
Sensitivity and specificity of BioFire FilmArray BCID2 Panel compared to conventional blood cultures in the subgroup of patients under antibiotic treatment or whom received antibiotic 48h before the febrile neutropenia onset. | 14 days
  * The sensitivity of the Biofire FilmArray BCID2 panel will be compared with the sensitivity of the companion blood cultures in the subgroup of patients with recent (<48 h) or concomitant use of systemic antibiotics. The results of the Biofire FilmArray samples that meet the definitions of "Proven BSI", "Probable BSI" and "Possible BSI" will be considered as positive results. The results will be assessed at Day 14 from the blood sample collection. The positive predictive value of both techniques will be calculated and compared.
  * The specificity of the Biofire FilmArray BCID2 panel will be compared with the specificity of the companion blood cultures in the subgroup of patients with recent (<48 h) or concomitant use of systemic antibiotics. The results will be assessed at Day 14 from the sample collection. The negative predictive value of both techniques will be calculated and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Carlota Gudiol, Professor, MD, PhD, Principal Investigator — Bellvitge University Hospital
Locations (1):
- Bellvitge University Hospital, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Patient´s age and sex, underlying disease and immunosuppressive therapies, clinical presentation, vital signs, duration of neutropenia, date of the initial blood cultures collection, cultures from other sites of infection collected within a time window of 10 days, blood count and chemistry, (including inflammatory biomarkers), and antimicrobial prescription (previous, current and posterior to the febrile neutropenia onset during study observation and 30 days before). Data regarding the microbiological results of the collected samples for each episode of febrile neutropenia will be collected. Date and time of febrile neutropenia episode, of blood cultures drawing and of blood cultures reception at Microbiology Laboratory will be registered. For both strategies microorganism identification, time to species identification, resistance mechanisms and time to resistance mechanism detection will be registered.
Supporting Information: Study Protocol
Time Frame: The study protocol is being written, and is planned to be published during the first six months of 2025
Access Criteria: The study protocol will be published in an Open access journal.

REFERENCES:
- [Derived] Bergas A, Lopez de Egea G, Albasanz-Puig A, Machado M, Vinado B, Estevez-Prieto A, Maluquer C, Carro I, Perez-Gonzalez A, Regalado-Artamendi I, Gomez-Centurion IA, Laporte-Amargos J, Sastre-Escola E, Badia-Tejero AM, Garcia P, Larrosa N, Munoz P, Berbel D, Ardanuy C, Carratala J, Gudiol C. Effectiveness of the BioFire FilmArray for the rapid detection of bloodstream infection in haematological patients with febrile neutropenia (the ONFIRE study): study protocol of a prospective, multicentre observational study at three reference university hospitals in Spain. BMJ Open. 2025 Jun 10;15(6):e101040. doi: 10.1136/bmjopen-2025-101040. PMID 40499967
- See also: BioFire FilmArray BCID2 panel manufacturer's instructions — https://www.biomerieux.com/us/en/our-offer/clinical-products/biofire-blood-culture-identification-2-panel.html